CLINICAL TRIAL: NCT00951340
Title: Desensitization and Cognitive Therapy in General Anxiety.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michelle G. Newman, Professor of Psychology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH039172-02 (NIH); R01MH039172-02 (NIH); 2R01MH039172-12 (NIH)
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Generalized Anxiety Disorder
Keywords: CBT; Emotional-Focused Therapy; Interpersonal Therapy
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Cognitive Behavioral Therapy; glutamate decarboxylase 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT with listening therapy (Active Comparator): Participants will receive CBT with listening therapy.
  Interventions: Other: Cognitive behavioral therapy (CBT); Behavioral: Listening therapy
- CBT with emotional processing and interpersonal therapy (Experimental): Participants will receive CBT with emotional processing and interpersonal therapy.
  Interventions: Other: Cognitive behavioral therapy (CBT); Behavioral: Emotional processing and interpersonal therapy

INTERVENTIONS:
Other: Cognitive behavioral therapy (CBT) — 15 weekly therapy sessions, the first hour of which will be devoted to standard CBT techniques
  Other Names: CBT for GAD
Behavioral: Emotional processing and interpersonal therapy — 15 weekly therapy sessions, the second hour of which will be devoted to interpersonal and emotional processing therapy techniques
  Arms: CBT with emotional processing and interpersonal therapy
Behavioral: Listening therapy — 15 weekly therapy sessions, the second hour of which will be directed by the participant's questions and discussion
  Arms: CBT with listening therapy

SUMMARY:
This study will test the feasibility and safety of adding interpersonal and emotional processing techniques to standard cognitive behavioral therapy for generalized anxiety disorder.

DETAILED DESCRIPTION:
Generalized anxiety disorder (GAD) is characterized by chronic worry that interrupts normal functioning. Some research has shown cognitive behavioral therapy (CBT) as an effective treatment for GAD, but only half of people treated with CBT for GAD experience treatment benefits long-term. Standard CBT for GAD may lose effectiveness over time because it does not address interpersonal and emotional processing problems. This study will determine the safety and feasibility of training therapists to deliver a version of CBT with additional therapeutic techniques for addressing interpersonal interactions and emotional processing.

Participation in this study will include 14 weekly, 2-hour, individual therapy sessions. During the first hour of each session, all participants will receive standard CBT for GAD. Participants will be randomly assigned to receive one of two therapies during the second hour: training in interpersonal and emotional processing techniques or listening therapy. Participants taking medications will be required to maintain a fixed dosage and keep a daily dairy of medication use, starting 2 weeks before study entry and lasting throughout treatment.

In-depth study assessments will take place at baseline and after completing the 15 weeks of therapy. Assessments will include clinical interviews, self-report questionnaires, and a physiological measurement session. Questions will pertain to anxiety symptoms, self-perceptions, emotional experience, and perceptions of the world. The physiological measurement session will involve recording bodily reactions, including brain waves, heart rate, eye movement, and breathing, while performing simple perceptual tasks. Brief psychological assessments will also follow each hour-long portion of each therapy session. Follow-up assessments conducted 6, 12, and 24 months after completing treatment will involve interviews and questionnaires as well as recording a week's worth of medication diaries.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of generalized anxiety disorder (GAD), as defined by the DSM-IV and agreed on by two diagnostic interviewers

Exclusion Criteria:

* Concurrent psychosocial therapy or past adequate dosage of CBT
* Medical contributions to anxiety
* Current substance abuse, psychosis, or organic brain syndrome

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 1996-07; Primary Completion 1998-07 (Actual); Study Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of delivering emotional processing and interpersonal therapeutic techniques | Measured at baseline, post-treatment, and after 6, 12, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michelle G. Newman, PhD, Study Director — Penn State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

REFERENCES:
- [Result] Newman MG, Castonguay LG, Borkovec TD, Fisher AJ, Nordberg SS. AN OPEN TRIAL OF INTEGRATIVE THERAPY FOR GENERALIZED ANXIETY DISORDER. Psychotherapy (Chic). 2008 Jun 1;45(2):135-147. doi: 10.1037/0033-3204.45.2.135. PMID 19881891